CLINICAL TRIAL: NCT01888952
Title: Phase 0/1 Biomarker and Pharmacodynamic Study of Roflumilast in Patients With Advanced B-Cell Hematologic Malignancies (CTRC# 13-0013)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anand B. Karnad (Other)
Responsible Party: Sponsor-Investigator, Anand B. Karnad, Principal Investigator, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRC 13-0013; HSC20130307H (Other: University of Texas Health Science Center San Antonio IRB (UTHSCSA))
Record Dates: First submitted 2013-05-08; First posted 2013-06-28 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Advanced B-cell Lymphoid Malignancies
MeSH Terms: interventions — Prednisone; Roflumilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Roflumilast and Prednisone (Experimental): Roflumilast 500 mcg will be administered orally daily for 21 consecutive days (a 21-day cycle).
  In Cycle 1, prednisone 60 mg/m2 up to a maximum of 100 mg oral (PO) daily will be taken on Days 8 through 14 at the same time as roflumilast.
  In Cycle 2 and subsequent cycles, prednisone 60 mg/m2 PO up to a maximum of 100 mg daily will be taken on Days 1 through 7 at the same time as roflumilast.
  Interventions: Drug: Prednisone; Drug: Roflumilast

INTERVENTIONS:
Drug: Prednisone — Patients may receive additional courses of treatment with prednisone (and roflumilast) at the discretion of the investigator if they did not experience unacceptable toxicity and have stable disease or objectively responding disease.
  Other Names: Deltasone
Drug: Roflumilast — Patients may receive additional courses of treatment with roflumilast (and prednisone) at the discretion of the investigator if they did not experience unacceptable toxicity, and have stable disease or objectively responding disease.
  Other Names: Daliresp

SUMMARY:
This is a Phase 0/1 open-label, non-randomized, biomarker and pharmacodynamic study in patients with advanced B-cell lymphoid malignancies, including B-cell chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), acute lymphocytic leukemia (ALL), multiple myeloma (MM), Waldenström's macroglobulinemia (WM), mantle cell lymphoma, follicular lymphoma, or diffuse large B-cell lymphoma (DLBCL) who have failed at least one prior therapy and for whom no standard curative therapy exists. Patients with advanced stage disease are those whose disease is resistant or refractory to standard chemotherapy or biological therapies.

DETAILED DESCRIPTION:
This pilot study will evaluate whether the administration of roflumilast inhibits the activity of PDE4 and results in the modulation of AKT/mTOR pathways in patients with B-cell hematologic malignancies. Peripheral blood samples will be collected for the purpose of determining the pharmacodynamics of roflumilast on PDE4 activity and on biomarkers as related to GC resistance. Samples are obtained at baseline prior to starting study treatment, on Day 8 before the administration of the Day 8 study drugs (prednisone and roflumilast), and on Day 15. If a bone marrow biopsy is also performed prior to study treatment or at any time during treatment, a sample will be sent for analysis. Normal PBMC (and bone marrow when it is obtained) will be examined for changes in key targets related to the inhibition of PDE4 and potential reversal of glucocorticoid resistance. Biomarker blood samples will be analyzed in order to characterize the pharmacodynamics of roflumilast alone and in combination with prednisone on PDE4 activity and on biomarkers, such as phospho-AKT, phosphorylation levels of mTOR targets.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Men and women > 18 years of age
* Diagnosed with relapsed or refractory (per investigator assessment) B-cell hematologic malignancy, including CLL, SLL, ALL, MM, WM, mantle cell lymphoma, follicular lymphoma, or DLBCL that has progressed or recurred following prior therapy. Patients must have failed, refused, be ineligible, or not otherwise appropriate for any potential standard curative treatment. In addition, patients must be refractory to or intolerant of established therapy known to provide clinical benefit for their condition. The original diagnostic biopsy and/or other diagnostic data (e.g., cell marker data) will suffice.
* Has failed ≥ 1 previous treatment for their malignancy, and has relapsed or refractory disease following most recent prior treatment.
* ECOG performance status of ≤ 2 and a life expectancy of at least 3 months.
* Ability to swallow oral tablets without difficulty.
* All subjects with preserved reproductive potential must agree to practice abstinence or employ contraceptive measures for the duration of treatment and for 4 weeks following final dosing.

  * All male subjects are considered to have reproductive potential.
  * Female subjects of reproductive potential are those who: 1) are not at least 50 years old and have no menses for 24 consecutive months; or 2) have not been rendered surgically sterile (having undergone hysterectomy and/or bilateral salpingo-oophorectomy).
  * Female subjects of reproductive potential must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin ([hCG]) within 7 days of first day of drug dosing.
* Has recovered from adverse, toxic effects of prior therapies to ≤ Grade 1(NCI-CTCAE v4) except for alopecia and peripheral neuropathy. This requirement will be subordinate to specific clinical and laboratory criteria that are otherwise specifically addressed in these inclusion/exclusion criteria. Peripheral neuropathy must have recovered to ≤ Grade 2 except for patients with WM, who may enroll with Grade 3 peripheral neuropathy if due to the underlying WM.
* Meet the following clinical laboratory requirements:

All patients, except ALL:

* Creatinine clearance by Cockcroft-Gault formula of ≥30 ml/min
* Total bilirubin ≤ 1.5 × ULN (unless indirect bilirubin is elevated due to Gilbert's syndrome or hemolysis)
* Aspartate aminotransaminase (AST) and alanine aminotransaminase (ALT) ≤ 3 × ULN
* Platelet count ≥ 50,000/uL, patients may be transfused to this value.
* Absolute neutrophil count (ANC) ≥ 1000/uL, with or without chronic granulocyte growth factor support
* Hemoglobin ≥8 g/dL, patients may be transfused to this value

For patients with ALL and CLL:

The hematological criteria do not apply.

Exclusion Criteria:

* Prior allogeneic bone marrow transplant within 6 months of screening date.
* Prior autologous stem cell transplant within 3 months of screening date.
* Active central nervous system (CNS) involvement by lymphoma, including untreated symptomatic epidural disease.
* Patients with autoimmune hemolytic anemia or immune thrombocytopenia requiring on-going active immunotherapy at study entry other than systemic corticosteroids less than or equal to prednisone equivalent 20 mg/day.
* Allergy or intolerance to roflumilast.
* Immunotherapy, chemotherapy, radiotherapy or investigational therapy within 3 weeks (within 4 weeks for monoclonal antibodies; within 6 weeks for nitrosoureas; within 12 weeks for iodine-131 tositumomab and ibritumomab tiuxetan) prior to study drug dosing.
* Active uncontrolled infection.
* Is receiving concurrent high doses of systemic corticosteroids. High dose is considered as >20 mg of dexamethasone a day (or equivalent) for >7 consecutive days.
* Uncontrolled illness including but not limited to: symptomatic congestive heart failure (New York Heart Association [NYHA] Class III or IV heart failure), unstable angina pectoris, uncontrolled cardiac arrhythmia, and psychiatric illness that would limit compliance with study requirements.
* History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty and/or stenting within 6 months prior to study drug dosing.
* History of another currently active cancer or any other cancer < 2 years prior to study drug dosing, except for adequately treated basal cell or squamous cell carcinoma of the skin, cervical cancer in situ or other adequately treated in situ carcinoma.
* Patients with a history of major surgery within 3 weeks or minor surgery within one week of roflumilast administration. Major surgery includes, for example, any open or laparoscopic entry into a body cavity, or operative repair of fracture; minor surgery includes, for example, open surgical biopsy of palpable/superficial lymph node, or placement of vascular access device.
* Other medical or psychiatric illness or organ dysfunction, which in the opinion of the investigator, would either compromise the subject's safety or interfere with the evaluation of the safety of the study agent.
* Corrected QT interval (QTc) prolongation (defined as a QTc >450 msec for males and >470 msec for females [Fridericia's correction]) or other clinically significant ECG abnormalities as assessed by the investigator.
* Patients known to be HIV-positive must not have multi-drug resistant HIV infection, CD4 counts < 150/mcl or other concurrent AIDS-defining conditions.
* Patients positive for Hepatitis B surface antigen (HBsAg) or Hepatitis C-virus ribonucleic acid (HCV RNA), unless both AST and ALT≤1.25 x ULN and no known history of chronic active hepatitis.
* Patients with moderate to severe liver impairment (Child-Pugh B or C)
* Women who are pregnant or breastfeeding.
* Patients with a history of depression or other psychiatric illness
* Patients who are taking strong cytochrome P450 enzyme inducers and inhibitors.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Karnad, MD, Principal Investigator — CTRC @ UTHSCSA; Ricardo Aguiar, MD PhD, Principal Investigator — CTRC @ UTHSCSA
Locations (1):
- Ctrc @ Uthscsa, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Roflumilast and Prednisone: Roflumilast 500 mcg will be administered orally daily for 21 consecutive days (a 21-day cycle).
  In Cycle 1, prednisone 60 mg/m2 up to a maximum of 100 mg oral (PO) daily will be taken on Days 8 through 14 at the same time as roflumilast.
  In Cycle 2 and subsequent cycles, prednisone 60 mg/m2 PO up to a maximum of 100 mg daily will be taken on Days 1 through 7 at the same time as roflumilast.
  Prednisone: Patients may receive additional courses of treatment with prednisone (and roflumilast) at the discretion of the investigator if they did not experience unacceptable toxicity and have stable disease or objectively responding disease.
  Roflumilast: Patients may receive additional courses of treatment with roflumilast (and prednisone) at the discretion of the investigator if they did not experience unacceptable toxicity, and have stable disease or objectively responding disease.
Period: Overall Study
Arm/Group | Roflumilast and Prednisone
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Roflumilast and Prednisone
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Adverse Events.
Description: Adverse events were listed using CTCAE Version 4.03 (Common Terminology Criteria for Adverse Events) toxicity grade.
Time Frame: Average of 21 days.
Measure: Number; unit: Adverse events
Arm/Group | Roflumilast and Prednisone
Number analyzed (Participants) | 10
Adverse events | 2

ADVERSE EVENTS:
Arm/Group | Roflumilast and Prednisone
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roflumilast and Prednisone (N=10)
Fatigue (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes